CLINICAL TRIAL: NCT04517916
Title: Zephyr Etude Post-Inscription (French Registry)
Status: Active, not recruiting | Type: Observational
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 630-0029-01
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Emphysema or COPD
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Zephyr Valve treatment: Patients undergoing the Zephyr Valve treatment for emphysema/COPD
  Interventions: Device: Zephyr Valve

INTERVENTIONS:
Device: Zephyr Valve — Subjects prescribed Zephyr Valve treatment for their emphysema/COPD and treated with the Zephyr Valves.
  Other Names: Zephyr System; BLVR

SUMMARY:
The objective of this Registry is to provide ongoing safety and effectiveness assessment of the Zephyr Valve treatment of adult patients with Chronic Obstructive Pulmonary Disease (COPD) Grade III and Grade IV in order to support the renewal of the inscription of the Zephyr Valve on the list LPPR (Art 165-1) in France.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, prospective Registry to be conducted at a minimum of 12 study centers. Approximately 150 patients with severe emphysema undergoing Zephyr Valve treatment will be enrolled and followed out to 3 years. Assessments will be performed at 45-days, 6-months, 12-months, 24-months and 36-months post-procedure.

Patients prescribed the Zephyr Valve treatment will be consented and will be enrolled only after determination of little to no collateral ventilation between target and ipsilateral lobes. Safety and effectiveness of the Zephyr Valve treatment will be evaluated post-treatment based on data collected out to 3-years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with emphysema (COPD Grade III and Grade IV) considered appropriate for the bronchoscopic lung volume reduction procedure by the physician.
* Subjects who signed an Informed Consent Form to allow data collection.

Exclusion Criteria:

* Subjects determined to have collateral ventilation between the target(s) and ipsilateral lobe(s).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is an all-comers Registry. Physicians at participating study centers will invite consecutive patients who are prescribed Zephyr Valve treatment to participate in the Registry and allow data collection.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 12 months
  The percent of patients achieving an improvement in the post-bronchodilator FEV1 of ≥12% at 12-months.

SECONDARY OUTCOMES:
Treated Lobar Volume Reduction (TLVR) | 45 days
  Treated Lobar Volume Reduction (TLVR) assessed by High Resolution Computed Tomography (HRCT) at 45-days.

OTHER OUTCOMES:
Absolute Change in Forced Expiratory Volume in 1 second FEV1 Post-Bronchodilator | Baseline, 6-months, 12-months, 24-months and 36-months
  Absolute Change in FEV1 from Baseline to 6-months, 12-months, 24-months and 36-months.
Percent Change in Forced Expiratory Volume in 1 second FEV1 Post-Bronchodilator | Baseline, 6-months, 12-months, 24-months and 36-months
  Percent change in FEV1 from Baseline to 6-months, 12-months, 24-months and 36-months.
Absolute Change in Residual Volume (RV) | Baseline, 6-months, 12-months, 24-months and 36-months
  Absolute Change in Residual Volume (RV) from Baseline to 6-months, 12-months, 24-months and 36-months.
Percent Change in Residual Volume (RV) | Baseline, 6-months, 12-months, 24-months and 36-months
  Percent change in Residual Volume (RV) from Baseline to 6-months, 12-months, 24-months and 36-months.
Absolute Change in St. George's Respiratory Questionnaire (SGRQ) Total Score | Baseline, 6-months and 12-months
  Absolute change in St. George's Respiratory Questionnaire (SGRQ) from Baseline to 6-months and 12-months.
  The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. Scores range from 0 to 100, with higher scores indicating more limitations.
Percent Change in St. George's Respiratory Questionnaire (SGRQ) Total Score | Baseline, 6-months and 12-months
  Percent change in St. George's Respiratory Questionnaire (SGRQ) Total Score from Baseline to 6-months and 12-months.
  The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. Scores range from 0 to 100, with higher scores indicating more limitations.
Absolute Change in Modified Medical Research Council (mMRC) | Baseline, 6-months and 12-months
  Absolute Change in the Modified Medical Research Council (mMRC) Dyspnea Scale from Baseline to 6-months and 12-months.
  The mMRC (Modified Medical Research Council) stratifies severity of dyspnea in respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4, with higher scores indicating more limitations.
Percent Change in Modified Medical Research Council (mMRC) | Baseline, 6-months and 12-months
  Percent change in the Modified Medical Research Council (mMRC) Dyspnea Scale from Baseline to 6-months and 12-months.
  The mMRC (Modified Medical Research Council) stratifies severity of dyspnea in respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4, with higher scores indicating more limitations.
Absolute Change in Six-Minute Walk Distance (6MWT) | Baseline, 6-months and 12-months.
  Absolute change in Six-Minute Walk Distance (from 6MWT) from Baseline to 6-months and 12-months.
Percent Change in Six-Minute Walk Distance (6MWT) | Baseline, 6-months and 12-months.
  Percent change in Six-Minute Walk Distance (from 6MWT) from Baseline to 6-months and 12-months.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Egenod, MD, Principal Investigator — Hôpital Dupuytren (CHRU Limoges); Dennis McHugh, Study Director — Pulmonx Corporation
Locations (12):
- France (12):
  - Hôpital La Cavale Blanche, Brest
  - Hôpital François Mitterrand, Dijon
  - Hôpital Nord, Latronche
  - Hôpital Calmette, Lille
  - Hôpital Dupuytren, Limoges
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Bichat, Paris
  - Hôpital Cochin, Paris
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Nord, Saint-Etienne
  - Nouvel Hôpital Civil, Strasbourg
  - Hôpital Larrey, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Criner GJ, Sue R, Wright S, Dransfield M, Rivas-Perez H, Wiese T, Sciurba FC, Shah PL, Wahidi MM, de Oliveira HG, Morrissey B, Cardoso PFG, Hays S, Majid A, Pastis N Jr, Kopas L, Vollenweider M, McFadden PM, Machuzak M, Hsia DW, Sung A, Jarad N, Kornaszewska M, Hazelrigg S, Krishna G, Armstrong B, Shargill NS, Slebos DJ; LIBERATE Study Group. A Multicenter Randomized Controlled Trial of Zephyr Endobronchial Valve Treatment in Heterogeneous Emphysema (LIBERATE). Am J Respir Crit Care Med. 2018 Nov 1;198(9):1151-1164. doi: 10.1164/rccm.201803-0590OC. PMID 29787288
- [Background] Kemp SV, Slebos DJ, Kirk A, Kornaszewska M, Carron K, Ek L, Broman G, Hillerdal G, Mal H, Pison C, Briault A, Downer N, Darwiche K, Rao J, Hubner RH, Ruwwe-Glosenkamp C, Trosini-Desert V, Eberhardt R, Herth FJ, Derom E, Malfait T, Shah PL, Garner JL, Ten Hacken NH, Fallouh H, Leroy S, Marquette CH; TRANSFORM Study Team *. A Multicenter Randomized Controlled Trial of Zephyr Endobronchial Valve Treatment in Heterogeneous Emphysema (TRANSFORM). Am J Respir Crit Care Med. 2017 Dec 15;196(12):1535-1543. doi: 10.1164/rccm.201707-1327OC. PMID 28885054
- [Background] Valipour A, Slebos DJ, Herth F, Darwiche K, Wagner M, Ficker JH, Petermann C, Hubner RH, Stanzel F, Eberhardt R; IMPACT Study Team. Endobronchial Valve Therapy in Patients with Homogeneous Emphysema. Results from the IMPACT Study. Am J Respir Crit Care Med. 2016 Nov 1;194(9):1073-1082. doi: 10.1164/rccm.201607-1383OC. PMID 27580428
- [Background] Klooster K, ten Hacken NH, Hartman JE, Kerstjens HA, van Rikxoort EM, Slebos DJ. Endobronchial Valves for Emphysema without Interlobar Collateral Ventilation. N Engl J Med. 2015 Dec 10;373(24):2325-35. doi: 10.1056/NEJMoa1507807. PMID 26650153
- [Background] Klooster K, Hartman JE, Ten Hacken NH, Slebos DJ. One-Year Follow-Up after Endobronchial Valve Treatment in Patients with Emphysema without Collateral Ventilation Treated in the STELVIO Trial. Respiration. 2017;93(2):112-121. doi: 10.1159/000453529. Epub 2016 Dec 15. PMID 27974713